CLINICAL TRIAL: NCT00461149
Title: Beneficial Effect of Dose Escalation of Octreotide-LAR as First-Line Therapy in Patients With Resistant Acromegaly
Brief Title: Dose Escalation of Octreotide-LAR as First-Line Therapy in Resistant Acromegaly
Acronym: HDacro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-1
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; GH; IGF-I; Pituitary tumors; Octreotide
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Octreotide-LAR

SUMMARY:
Epidemiological data indicate that patients with active acromegaly have reduced life expectancy because of cardiovascular (60%) and respiratory diseases (25%) mainly (1-10). A post-treatment GH value <5 mU/liter (equal to <2.5 μg/liter) and IGF-I in the normal range for age are recognized as the most predictive survival indices.

Since their introduction into clinical use approximately two decades ago, somatostatin analogs have been considered a cornerstone of medical therapy for acromegaly. After 12 months of treatment with octreotide-LAR, control of GH and IGF-I excess, is achieved in 54% and 63% of unselected patients (11). The proportion of subjects achieving IGF-I normalization increases significantly with time (12). Significant tumor shrinkage has also been reported in a number of studies (13,14): an average 50% tumor decrease is achieved when the drug is used exclusively, or before surgery or radiotherapy (14). In 99 unselected newly diagnosed patients after 12 months of treatment with somatostatin analogues we reported control of GH levels in 57.6% and IGF-I levels in 45.5% and a greater than 50% tumor shrinkage in 44.4% (15).

The dose of LAR in different studies ranged from 10-40 mg every 28 days (q28d): high doses are generally administered in patients who do not control GH and IGF-I excess with lower doses. As reported in the meta-analysis (11) the rate of IGF-I normalization tended to be lower as octreotide-LAR dose was raised: 90% in patients treated with 10 mg, 61% with 20 mg and 53% with 30 mg. However, some further benefit by increasing the dose of octreotide-LAR was reported in some studies (16-18).

Data on dose escalation of octreotide-LAR given as first-line therapy in newly diagnosed patients with acromegaly are lacking.

DETAILED DESCRIPTION:
This is an analytical, interventional, 24-month, open, prospective study to investigate the effect of progressive increase of octreotide-LAR doses in newly diagnosed patients with acromegaly. Primary outcome measures were GH and IGF-I control and tumor shrinkage; secondary outcome measure was glucose tolerance.

At diagnosis and every six months, 24-48 hours before changes in treatment doses was applied, were measured:

1. Serum IGF-I levels twice in a single sample at the time 0 of the GH profile; GH levels calculated as the mean value of 3-6 samples drawn every 30 min; the average value was considered for the statistical analysis;
2. Tumor volume on MRI studies performed on clinical 1T and 1.5T scanners, using T1 weighted gradient recalled-echo in the sagittal and coronal planes, as already reported (15,21,22). The acquisitions were repeated before and after the administration of 0.1 mmoles of gadolinium chelate (diethylene-triamine pentacetate). In all patients MRI was performed at diagnosis and after 6, 12, and 24 months of treatment. The maximal sagittal, axial and coronal diameters were measured, then tumor volume was calculated by the De Chiro and Nelson formula [(volume= sagittal*coronal*axial diameters)*π/6]. According with previous studies (13,21) on post-treatment MRI, tumor shrinkage was assessed as percent decrease of tumor volume compared with baseline.
3. Glucose tolerance by assaying glucose and insulin levels at fasting. Only at diagnosis glucose and insulin were also measured every 30 minutes for 2 hours after the oral administration of 75 g of glucose diluted in 250 ml of saline solution. In four patients the glucose load was not performed because of overt diabetes (fasting glucose was above 7 mmol/L at two consecutive measurements) (25). Diabetes mellitus was diagnosed in another eight patients when 2 hours after the oGTT glucose was >11 mmol/L (25). Impaired glucose tolerance (IGT) when glucose level was between >7.8 mmol/L and <11 mmol/L 2 hours after the oGTT and/or impaired fasting glucose (IFG) when glucose level was between 5.6 and 6.9 mmol/L at fasting were diagnosed in 20 patients (25). Glucose tolerance was normal (below 5.6 mmol/L at fasting) in 24 patients. To predict insulin resistance [HOMA-R (%)] and ß-cell function [HOMA-β (%)] was used the HOMA (homeostatic model assessment) according with Matthews et al. (24). By assuming that normal-weight healthy subjects aged <35 years have a HOMA-β of 100% and a HOMA-R of 1, the values for individual patients can be assessed from the insulin and glucose concentrations by the formulae: HOMA-R = [insulin (mU/L)*fasting glucose (mmol/L)] / 22.5; HOMA-β (%) = [20*insulin (mU/L)] / [glucose (mmol/L)-3.5].

Treatment protocol Before starting therapy, all patients received an acute test with s.c. octreotide at a dose of 0.1 mg in the morning after an overnight fast and at least 2 hrs of bedrest, to investigate each patient's tolerability to somatostatin analogues (25). Then, all patients were treated with octreotide-LAR i.m. at an initial dose of 20 mg every 28 days for three months. Subsequently, LAR treatment was maintained at the same dose in patients achieving GH levels ≤2.5 μg/liter and IGF-I levels in the normal range (Group A), or increased up to 30 mg every 28 days in patients with GH levels >2.5 μg/liter and/or IGF-I levels above the normal range. After another 9 months of treatment with 30 mg/q28d, the dose was maintained in 15 patients achieving GH levels ≤2.5 μg/liter and IGF-I levels in the normal range (Group B) while it was further increased to 40 mg/q28 days if fasting GH levels were still >2.5 μg/liter and/or IGF-I levels were above the normal range (Group C).

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed acromegaly
* age above 18 years
* no previous treatments for acromegaly

Exclusion Criteria:

* primary surgery
* concomitant hyperprolactinemia if requiring combined treatment with dopamine-agonist
* primary treatment with lanreotide
* treatment duration less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1995-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
GH and IGF-I control
tumor shrinkage

SECONDARY OUTCOMES:
Glucose tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria AL Colao, Prof., Principal Investigator — University Federico II
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology University Federico II of Naples, Naples, Italy

REFERENCES:
- [Result] Wright AD, Hill DM, Lowy C, Fraser TR. Mortality in acromegaly. Q J Med. 1970 Jan;39(153):1-16. No abstract available. PMID 5427331
- [Result] Bates AS, Van't Hoff W, Jones JM, Clayton RN. An audit of outcome of treatment in acromegaly. Q J Med. 1993 May;86(5):293-9. PMID 8327647
- [Result] Etxabe J, Gaztambide S, Latorre P, Vazquez JA. Acromegaly: an epidemiological study. J Endocrinol Invest. 1993 Mar;16(3):181-7. doi: 10.1007/BF03344942. PMID 8514973
- [Result] Rajasoorya C, Holdaway IM, Wrightson P, Scott DJ, Ibbertson HK. Determinants of clinical outcome and survival in acromegaly. Clin Endocrinol (Oxf). 1994 Jul;41(1):95-102. doi: 10.1111/j.1365-2265.1994.tb03789.x. PMID 8050136
- [Result] Abosch A, Tyrrell JB, Lamborn KR, Hannegan LT, Applebury CB, Wilson CB. Transsphenoidal microsurgery for growth hormone-secreting pituitary adenomas: initial outcome and long-term results. J Clin Endocrinol Metab. 1998 Oct;83(10):3411-8. doi: 10.1210/jcem.83.10.5111. PMID 9768640
- [Result] Swearingen B, Barker FG 2nd, Katznelson L, Biller BM, Grinspoon S, Klibanski A, Moayeri N, Black PM, Zervas NT. Long-term mortality after transsphenoidal surgery and adjunctive therapy for acromegaly. J Clin Endocrinol Metab. 1998 Oct;83(10):3419-26. doi: 10.1210/jcem.83.10.5222. PMID 9768641
- [Result] Orme SM, McNally RJ, Cartwright RA, Belchetz PE. Mortality and cancer incidence in acromegaly: a retrospective cohort study. United Kingdom Acromegaly Study Group. J Clin Endocrinol Metab. 1998 Aug;83(8):2730-4. doi: 10.1210/jcem.83.8.5007. PMID 9709939
- [Result] Ayuk J, Clayton RN, Holder G, Sheppard MC, Stewart PM, Bates AS. Growth hormone and pituitary radiotherapy, but not serum insulin-like growth factor-I concentrations, predict excess mortality in patients with acromegaly. J Clin Endocrinol Metab. 2004 Apr;89(4):1613-7. doi: 10.1210/jc.2003-031584. PMID 15070920
- [Result] Holdaway IM, Rajasoorya RC, Gamble GD. Factors influencing mortality in acromegaly. J Clin Endocrinol Metab. 2004 Feb;89(2):667-74. doi: 10.1210/jc.2003-031199. PMID 14764779
- [Result] Kauppinen-Makelin R, Sane T, Reunanen A, Valimaki MJ, Niskanen L, Markkanen H, Loyttyniemi E, Ebeling T, Jaatinen P, Laine H, Nuutila P, Salmela P, Salmi J, Stenman UH, Viikari J, Voutilainen E. A nationwide survey of mortality in acromegaly. J Clin Endocrinol Metab. 2005 Jul;90(7):4081-6. doi: 10.1210/jc.2004-1381. Epub 2005 May 10. PMID 15886256
- [Result] Freda PU, Katznelson L, van der Lely AJ, Reyes CM, Zhao S, Rabinowitz D. Long-acting somatostatin analog therapy of acromegaly: a meta-analysis. J Clin Endocrinol Metab. 2005 Aug;90(8):4465-73. doi: 10.1210/jc.2005-0260. Epub 2005 May 10. PMID 15886238
- [Result] Cozzi R, Montini M, Attanasio R, Albizzi M, Lasio G, Lodrini S, Doneda P, Cortesi L, Pagani G. Primary treatment of acromegaly with octreotide LAR: a long-term (up to nine years) prospective study of its efficacy in the control of disease activity and tumor shrinkage. J Clin Endocrinol Metab. 2006 Apr;91(4):1397-403. doi: 10.1210/jc.2005-2347. Epub 2006 Jan 31. PMID 16449332
- [Result] Bevan JS. Clinical review: The antitumoral effects of somatostatin analog therapy in acromegaly. J Clin Endocrinol Metab. 2005 Mar;90(3):1856-63. doi: 10.1210/jc.2004-1093. Epub 2004 Dec 21. PMID 15613435
- [Result] Melmed S, Sternberg R, Cook D, Klibanski A, Chanson P, Bonert V, Vance ML, Rhew D, Kleinberg D, Barkan A. A critical analysis of pituitary tumor shrinkage during primary medical therapy in acromegaly. J Clin Endocrinol Metab. 2005 Jul;90(7):4405-10. doi: 10.1210/jc.2004-2466. Epub 2005 Apr 12. PMID 15827109
- [Result] Colao A, Pivonello R, Auriemma RS, Briganti F, Galdiero M, Tortora F, Caranci F, Cirillo S, Lombardi G. Predictors of tumor shrinkage after primary therapy with somatostatin analogs in acromegaly: a prospective study in 99 patients. J Clin Endocrinol Metab. 2006 Jun;91(6):2112-8. doi: 10.1210/jc.2005-2110. Epub 2006 Mar 14. PMID 16537687
- [Result] Turner HE, Vadivale A, Keenan J, Wass JA. A comparison of lanreotide and octreotide LAR for treatment of acromegaly. Clin Endocrinol (Oxf). 1999 Sep;51(3):275-80. doi: 10.1046/j.1365-2265.1999.00853.x. PMID 10469005
- [Result] Cozzi R, Attanasio R, Montini M, Pagani G, Lasio G, Lodrini S, Barausse M, Albizzi M, Dallabonzana D, Pedroncelli AM. Four-year treatment with octreotide-long-acting repeatable in 110 acromegalic patients: predictive value of short-term results? J Clin Endocrinol Metab. 2003 Jul;88(7):3090-8. doi: 10.1210/jc.2003-030110. PMID 12843148
- [Result] Colao A, Ferone D, Marzullo P, Cappabianca P, Cirillo S, Boerlin V, Lancranjan I, Lombardi G. Long-term effects of depot long-acting somatostatin analog octreotide on hormone levels and tumor mass in acromegaly. J Clin Endocrinol Metab. 2001 Jun;86(6):2779-86. doi: 10.1210/jcem.86.6.7556. PMID 11397887
- [Result] Colao A, Lombardi G. Growth-hormone and prolactin excess. Lancet. 1998 Oct 31;352(9138):1455-61. doi: 10.1016/S0140-6736(98)03356-X. PMID 9808008
- [Result] Giustina A, Barkan A, Casanueva FF, Cavagnini F, Frohman L, Ho K, Veldhuis J, Wass J, Von Werder K, Melmed S. Criteria for cure of acromegaly: a consensus statement. J Clin Endocrinol Metab. 2000 Feb;85(2):526-9. doi: 10.1210/jcem.85.2.6363. PMID 10690849
- [Result] Colao A, Marzullo P, Ferone D, Spinelli L, Cuocolo A, Bonaduce D, Salvatore M, Boerlin V, Lancranjan I, Lombardi G. Cardiovascular effects of depot long-acting somatostatin analog Sandostatin LAR in acromegaly. J Clin Endocrinol Metab. 2000 Sep;85(9):3132-40. doi: 10.1210/jcem.85.9.6782. PMID 10999798
- [Result] Colao A, Pivonello R, Rosato F, Tita P, De Menis E, Barreca A, Ferrara R, Mainini F, Arosio M, Lombardi G. First-line octreotide-LAR therapy induces tumour shrinkage and controls hormone excess in patients with acromegaly: results from an open, prospective, multicentre trial. Clin Endocrinol (Oxf). 2006 Mar;64(3):342-51. doi: 10.1111/j.1365-2265.2006.02467.x. PMID 16487447
- [Result] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2006 Jan;29 Suppl 1:S43-8. No abstract available. PMID 16373932
- [Result] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Derived] Colao A, Pivonello R, Auriemma RS, Galdiero M, Savastano S, Lombardi G. Beneficial effect of dose escalation of octreotide-LAR as first-line therapy in patients with acromegaly. Eur J Endocrinol. 2007 Nov;157(5):579-87. doi: 10.1530/EJE-07-0383. PMID 17984237